CLINICAL TRIAL: NCT01403610
Title: A Phase 2, Investigator Initiated Study to Determine the Safety, Efficacy and CNS Penetration of TH-302 in Recurrent High Grade Astrocytoma Following Bevacizumab
Brief Title: Safety and Efficacy Study of TH-302 CNS Penetration in Recurrent High Grade Astrocytoma Following Bevacizumab
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: CTRC 11-24; CTRC 11-24 (Other: The Cancer Therapy and Research Center (CTRC))
Record Dates: First submitted 2011-07-22; First posted 2011-07-27 (Estimated); Results first posted 2019-07-24 (Actual); Last update posted 2019-07-24 (Actual); Status verified 2019-03

CONDITIONS: HIGH GRADE GLIOMA
Keywords: TH-302; Bevacizumab; Phase 2; Glioma; High Grade Glioma; CNS
MeSH Terms: conditions — Glioma | interventions — Drug Evaluation; TH 302

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Cohort 1 (Experimental): Subjects received TH-302 single dose at 575 mg/m2 or placebo administered preoperative in a 2:1 randomization and were then administered 240 mg/m2 of TH-302 post-operative.
  Interventions: Drug: TH-302 preoperative; Drug: Placebo; Drug: TH-302 (escalating) with bevacizumab 10mg/kg
- Cohort 2 (Experimental): Surgical subjects will receive TH-302 at 340 mg/m2 every 2 weeks (4 week cycles) starting after surgery from Cycle 1, Day 1 until disease progression.
  Interventions: Drug: TH-302 preoperative; Drug: TH-302 (escalating) with bevacizumab 10mg/kg
- Cohort 3 (Experimental): Surgical or Non-Surgical subjects will receive TH-302 at 480 mg/m2 every 2 weeks (4 week cycles) starting after surgery from Cycle 1, Day 1 until disease progression.
  Interventions: Drug: TH-302 (escalating) with bevacizumab 10mg/kg
- Cohort 4 (Experimental): Non-surgical subjects will receive a dose up to 670 mg/m2 of TH-302
  Interventions: Drug: TH-302 (escalating) with bevacizumab 10mg/kg

INTERVENTIONS:
Drug: TH-302 preoperative — TH-302 single dose at 575 mg/m2 administered preoperatively, followed by postoperative combination therapy bevacizumab at 10mg/kg every 2 weeks and TH-302 at 240 - 480 mg/m2 every 2 weeks (4 week cycle) until disease progression. Subjects will be randomized (2:1) to receive pre-operative dose of TH-302.
  Other Names: Study drug
  Arms: Cohort 1; Cohort 2
Drug: Placebo — Placebo administered preoperatively, followed by postoperative combination therapy bevacizumab at 10mg/kg every 2 weeks and TH-302 at 240 - 480 mg/m2 every 2 weeks (4 week cycle) until disease progression. Subjects will be randomized (2:1) to receive pre-operative dose of TH-302.
  Other Names: Study placebo
  Arms: Cohort 1
Drug: TH-302 (escalating) with bevacizumab 10mg/kg — Combination of 10mg/m2 of bevacizumab with an escalating dose of TH-302 from 240 to 670 mg/m2
  Other Names: Study drug escalating dose

SUMMARY:
The Primary Objectives are:

* To determine the extent by which TH-302 is able to penetrate the blood brain barrier and affect tumor tissue
* To assess the safety of single dose TH-302 in patients with high grade glioma undergoing surgery
* To assess the safety of TH-302 in combination with bevacizumab for patients with high grade glioma
* To determine the MTD and DLT(s) of TH-302 in combination with bevacizumab

The Secondary Objectives are:

To determine the progression-free survival with or without debulking craniotomy for patients treated with combination bevacizumab and TH-302 following recurrence on single agent bevacizumab

DETAILED DESCRIPTION:
Single center, dose-escalation, prospective study with TH-302 single dose at 575 mg/m2 or placebo administered preoperatively, followed by postoperative combination therapy bevacizumab at 10mg/kg every 2 weeks and TH-302 at 240 - 670 mg/m2 every 2 weeks (4 week cycle) until disease progression. Subjects will be randomized (2:1) to receive pre-operative dose of TH-302 (surgical subjects only). Subjects not receiving surgery will receive combination therapy of bevacizumab at 10 mg/kg every 2 weeks and TH-302 at 240-670 mg/m2 every 2 weeks (4 week cycle) starting from Cycle 1, Day 1 until disease progression.

This study will use a classic dose escalation design to determine the MTD of TH-302 when used in combination with bevacizumab. The dose of TH-302 will be escalated in cohorts of 3-6 subjects. The initial dose of TH-302 will be 240 mg/m2. A dose level minus 1 will be built into the study in the event that subjects experience excessive toxicity at Dose Level 1. Dose escalation will continue to 340 mg/m2 and 670 mg/m2.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age
2. Ability to understand the purposes and risks of the study and has signed a written informed consent form approved by the investigator's IRB/Ethics Committee
3. Histologically confirmed high grade astrocytoma
4. Progression following both standard combined modality treatment with radiation and temozolomide chemotherapy, as well as anti-angiogenic therapy (ie, bevacizumab)
5. Recovered from toxicities of prior therapy to grade 0 or 1
6. ECOG performance status of 0 or 1
7. Life expectancy of at least 3 months
8. Acceptable liver function
9. Acceptable renal function
10. Acceptable hematologic status
11. All women of childbearing potential must have a negative serum pregnancy test and male and female subjects must agree to use effective means of contraception (surgical sterilization or the use or barrier contraception with either a condom or diaphragm in conjunction with spermicidal gel or an IUD) with their partner from entry into the study through 6 months after the last dose

Exclusion Criteria:

1. The subject is receiving warfarin (or other coumarin derivatives) and is unable to switch to low molecular weight heparin (LMWH) before the first dose of study drug.
2. The subject has evidence of acute intracranial or intratumoral hemorrhage either by MRI or computerized tomography (CT) scan. Subjects with resolving hemorrhage changes, punctate hemorrhage, or hemosiderin are eligible.
3. The subject is unable to undergo MRI scan (eg, has pacemaker).
4. The subject has received enzyme-inducing anti-epileptic agents within 14 days of study drug (eg, carbamazepine, phenytoin, phenobarbital, primidone).
5. The subject has not recovered to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v4.0 Grade ≤ 1 from AEs (except alopecia, anemia and lymphopenia) due to surgery, antineoplastic agents, investigational drugs, or other medications that were administered prior to study drug.
6. The subject has evidence of wound dehiscence
7. Severe chronic obstructive or other pulmonary disease with hypoxemia (requires supplementary oxygen, symptoms due to hypoxemia or oxygen saturation <90% by pulse oximetry after a 2 minute walk) or in the opinion of the investigator any physiological state likely to cause normal tissue hypoxia
8. The subject is pregnant or breast-feeding.
9. The subject has serious intercurrent illness
10. The subject has inherited bleeding diathesis or coagulopathy with the risk of bleeding.
11. The subject has received any of the following prior anticancer therapy:

    * Non-standard radiation therapy such as brachytherapy, systemic radioisotope therapy (RIT), or intra-operative radiotherapy (IORT). Note: stereotactic radiosurgery (SRS) is allowed
    * Antiangiogenic agents whose primary mode of action is through the VEGF signaling within 21 days prior to first dose of study drug (surgical subjects only)
    * Non-bevacizumab systemic therapy (including investigational agents and small-molecule kinase inhibitors) or non-cytotoxic hormonal therapy (eg, tamoxifen) within 7 days or 5 half-lives, whichever is shorter, prior first dose of study drug
    * Biologic agents (antibodies, immune modulators, vaccines, cytokines) within 21 days prior to first dose of study drug
    * Nitrosoureas or mitomycin C within 42 days, or metronomic/protracted low-dose chemotherapy within 14 days, or other cytotoxic chemotherapy within 28 days, prior to first dose of study drug
    * Prior treatment with carmustine wafers
    * Prior treatment with TH-302

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2011-06; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Brenner, MD,, Principal Investigator — Institute for Drug Development
Locations (1):
- Cancer Therapy & Research Center at UTHSCSA, San Antonio, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: Prior to surgery subjects will be assigned to this group in a 2:1 randomization, ie. 2 subjects will be assigned to TH-302 and one to placebo. A single dose of 575 mg/m2 or placebo will be administered pre-operatively with hypoxyprobe-1 at 500 mg/m2 over 20 minutes. Subjects in this group receive TH-302 at a dose of 240mg/m2 post surgery.
- Cohort 2: Subjects received 340mg/m2 of TH-302 post surgery
- Cohort 3: Subjects were dosed with 480mg/m2 of TH-302 regardless of whether or not surgery was performed. 3 subjects in this arm had surgery prior to this dose of TH-302.
- Cohort 4: Subjects in this cohort did not undergo any surgery, a dose of 670mg/m2 was administered to all.
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Started | 5 | 6 | 4 | 13
Completed | 3 | 3 | 4 | 13
Not Completed | 2 | 3 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 0 | 0
Not completed — Didn't recover from surgery sufficiently | 0 | 3 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Total
Number analyzed (Participants) | 3 | 3 | 4 | 13 | 23
Age, Continuous [Mean (Full Range); unit: Years] | 56 [43 to 70] | 47 [44 to 51] | 50 [35 to 58] | 61 [42 to 74] | 56 [35 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3 | 3 | 9
  Male | 2 | 1 | 1 | 10 | 14
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 4 | 13 | 23

OUTCOME MEASURES:

1. Primary Outcome: Time to Progression
Description: Time from initiation study until radiographic progression by RANO criteria
Time Frame: 2 years
Population: See full published data at https://www.ncbi.nlm.nih.gov/pmc/articles/PMC6071657/
Measure: Median (Full Range); unit: months
Groups:
- Cohort 1: Bevacizumab (Bev) 10mg/kg every 2 weeks plus TH-302 240mg/m2 every 2 weeks (in a 4 week cycle)
- Cohort 2: Bevacizumab (Bev) 10mg/kg every 2 weeks plus TH-302 340mg/m2 every 2 weeks (in a 4 week cycle)
- Cohort 3: Bevacizumab (Bev) 10mg/kg every 2 weeks plus TH-302 480 mg/m2 every 2 weeks (in a 4 week cycle)
- Cohort 4: Bevacizumab (Bev) 10mg/kg every 2 weeks plus TH-302 470 mg/m2 every 2 weeks (in a 4 week cycle)
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 3 | 3 | 4 | 13
months | 11.3 [2.7 to 14] | 9 [7.8 to 14] | 15.6 [4.5 to 20] | 4.5 [1.8 to 14]

ADVERSE EVENTS:
Time Frame: 2 years
Description: Common Terminology Criteria for Adverse Events version 4.0, Grade 3 or higher reported as serious adverse events.
  Grade 1: Mild; asymptomatic or mild symptoms 2: Moderate; minimal, local or noninvasive intervention indicated 3: Severe or medically significant but not immediately life threatening 4: Life-threatening consequences; urgent intervention indicated. 5: Death
Groups:
- Cohort 1: 240 mg/m2 dosage
- Cohort 2: 340 mg/m2 dosage
- Cohort 3: 480 mg/m2 dosage
- Cohort 4: 670 mg/m2
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/4 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/3 | 1/3 | 1/4 | 0/13
Other Adverse Events (participants affected / at risk) | 1/3 | 2/3 | 1/4 | 7/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=3) | Cohort 2 (N=3) | Cohort 3 (N=4) | Cohort 4 (N=13)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=3) | Cohort 2 (N=3) | Cohort 3 (N=4) | Cohort 4 (N=13)
rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
anal inflammation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
proctitis (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hypertension (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No